CLINICAL TRIAL: NCT04603599
Title: Relationship of Endometrial Cancer and Serum Soluble L1CAM Level
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Merve Dermir, Director, Kocaeli University
Other Study IDs: Merve L1CAM
Record Dates: First submitted 2020-10-14; First posted 2020-10-27 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Endometrium Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- benign endometrial changes
  Interventions: Diagnostic Test: serum soluble L1CAM (sL1CAM)
- endometrial hyperplasia
  Interventions: Diagnostic Test: serum soluble L1CAM (sL1CAM)
- endometrial cancer
  Interventions: Diagnostic Test: serum soluble L1CAM (sL1CAM)

INTERVENTIONS:
Diagnostic Test: serum soluble L1CAM (sL1CAM) — blood sample

SUMMARY:
The aim of this study is to evaluate the effect of serum soluble L1CAM (sL1CAM) on the diagnosis and prognosis of endometrial cancer. This prospective randomized controlled trial will be conducted in patients who have undergone endometrial biopsy and whose pathology results are reported as benign endometrial changes, endometrial hyperplasia, or endometrial cancer. The sL1CAM level between groups will be compared. The relationship between prognostic factors and serum sL1CAM will be evaluated in patients with endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent endometrial biopsy due to abnormal uterine bleeding and whose pathology results were reported as benign endometrial changes, endometrial hyperplasia or endometrial cancer were included in the study. All patients participating in the study signed informed consent.

Exclusion Criteria:

* Patients who did not have consent, received neoadjuvant therapy and who would not have surgery despite endometrial cancer were excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: benign endometrial changes, endometrial hyperplasia or endometrial cancer
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
serum sL1CAM level | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Merve Demir, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided